CLINICAL TRIAL: NCT03400449
Title: Video Versus Conversational Contraceptive Counseling During Maternity Hospitalization: The COMSE Randomized Trial
Brief Title: Video Versus Conversational Contraceptive Counseling During Maternity Hospitalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Maureen Baldwin, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11331b
Record Dates: First submitted 2017-12-20; First posted 2018-01-17 (Actual); Results first posted 2019-06-19 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Contraceptive Usage; Contraception Behavior
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Intervention Model Description: Two groups randomized to counseling type.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video counseling (Active Comparator): The video group watched a 13.75 minute video of a local Colombian counselor reading a script of the same information provided by conversational counseling and had a chance to ask questions at the end.
  Interventions: Other: Video counseling
- Conversational counseling (Active Comparator): The conversation group participated in a structured, face-to-face conversation with a trained counselor.
  Interventions: Other: Conversational counseling

INTERVENTIONS:
Other: Video counseling — Video counseling
  Arms: Video counseling
Other: Conversational counseling — Conversational counseling
  Arms: Conversational counseling

SUMMARY:
A randomized trial comparing LARC uptake and satisfaction after either video or conversational-based contraceptive counseling for pregnant women in labor.

DETAILED DESCRIPTION:
This was a multi-center randomized, controlled trial examining contraceptive counseling in the setting of long-acting reversible contraception (LARC) uptake and immediate provision. At two urban public hospitals with large adolescent populations, participants were randomized to a structured, in-person conversation with a trained counselor or a 14-minute video providing the same information. Both participant groups were provided written materials and both had the opportunity to ask questions of the counselor. The total time to complete counseling was measured, as well as participant satisfaction, pre- and post-intervention contraceptive knowledge, and intended postpartum contraceptive method.

ELIGIBILITY:
Inclusion Criteria:

* Live pregnancy >20 weeks gestation
* Admission to maternity ward for labor
* Age >14

Exclusion Criteria:

* Pain >=8 on Wong-Baker FACES pain scale

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 240 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2016-08-07 (Actual); Study Completion 2016-08-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Colombia (2):
  - Maternidad Rafael Calvo, Cartagena
  - Metrosalud Manrique, Medellín

IPD SHARING:
Plan to Share IPD: No
Individual sites hold the paper data under monitoring plan through their site Institutional Review Board (IRB - University de Antioquia). They entered de-identified data electronically into REDCap for our use for analysis. We have shared aggregate analysis with the individual sites.

REFERENCES:
- [Derived] Hersh AR, Munoz LF, Rincon M, Alvarez C, Tolosa JE, Moreno DJ, Rubio M, Vargas JC, Edna F, Taborda N, Baldwin MK. Video compared to conversational contraceptive counseling during labor and maternity hospitalization in Colombia: A randomized trial. Contraception. 2018 Sep;98(3):210-214. doi: 10.1016/j.contraception.2018.05.004. Epub 2018 May 9. PMID 29752923

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Video Counseling | Conversational Counseling
Started | 121 | 119
Completed | 120 | 119
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Video Counseling | Conversational Counseling | Total
Number analyzed (Participants) | 120 | 119 | 239
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 23 | 43
  Between 18 and 65 years | 100 | 96 | 196
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 119 | 239
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Colombia | 120 | 119 | 239

OUTCOME MEASURES:

1. Primary Outcome: Total Counseling Time
Description: Duration of counseling in minutes (from initiation of counseling to conclusion of all questions answered.) The clock was not stopped for breaks, which were allowed as needed.
Time Frame: Immediately following the intervention, an average of less than 30 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Video Counseling | Conversational Counseling
Number analyzed (Participants) | 120 | 119
minutes | 16.8 (4.6) | 16.3 (4.6)

2. Secondary Outcome: Knowledge Scores
Description: Mean total correct answer (score) to 7 multiple-choice contraceptive knowledge questions. Total possible score is 0-7, with 7 representing 100% correct answers. Score measured after completion of the knowledge questionnaire, on average less than one hour, before (pre) and after (post) counseling.
Time Frame: One hour
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conversational Counseling | Video Counseling
Number analyzed (Participants) | 119 | 120
score on a scale
  Pre-counseling | 3.1 (1.5) | 3.1 (1.5)
  Post-counseling | 5.3 (1.0) | 5.1 (1.2)

3. Secondary Outcome: Number of Participants Initiating Postpartum LARC Uptake
Description: Number of participants initiating long-acting reversible contraception (LARC - intrauterine device (IUD) or implant) prior to hospital discharge.
Time Frame: Assessed at the time of hospital discharge, on average less than 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Conversational Counseling | Video Counseling
Number analyzed (Participants) | 119 | 120
Participants | 46 | 44

ADVERSE EVENTS:
Arm/Group | Video Counseling | Conversational Counseling
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/119
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/119
Other Adverse Events (participants affected / at risk) | 0/120 | 0/119

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No